CLINICAL TRIAL: NCT06580938
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION AND DOSE EXPANSION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND ANTI-TUMOR ACTIVITY OF PF-07921585 AS A SINGLE AGENT AND IN COMBINATION THERAPY IN PARTICIPANTS 18 YEARS OF AGE AND OLDER WITH ADVANCED SOLID TUMORS
Brief Title: A Study to Learn About PF-07921585 Alone or With Other Anti-cancer Medicines in People With Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated for strategic reasons. The decision was not based on any safety and/or efficacy concerns
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5461001; NCT06580938 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-08-05; First posted 2024-08-30 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer; Bladder Cancer; Renal Cell Carcinoma; Melanoma; Head and Neck Cancer; Colorectal Cancer
Keywords: Interleukin-12 mutein; Sasanlimab; anti-PD1 antibody; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Melanoma; Head and Neck Neoplasms; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Dose escalation monotherapy
  Interventions: Biological: PF-07921585
- Part 2 (Experimental): Dose escalation (combination therapy)
  Interventions: Biological: PF-07921585; Biological: Sasanlimab
- Part 3 (Experimental): Dose optimization/ expansion (combination therapy)
  Interventions: Biological: PF-07921585; Biological: Sasanlimab

INTERVENTIONS:
Biological: PF-07921585 — IL-12 mutein, solution, administered once every 3 weeks intravenously or subcutaneously
Biological: Sasanlimab — Anti-PD1 antibody solution, administered once every 3 weeks subcutaneously
  Other Names: PF-06801591
  Arms: Part 2; Part 3

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called PF-07921585) in people with cancer that has advanced or spread to other parts of the body.

This study is seeking participants who have any of the following cancer types:

* non-small cell lung cancer
* colorectal cancer
* bladder cancer
* melanoma (a type of skin cancer)
* kidney cancer
* head and neck cancer Participants will receive the study medicine PF-07921585 alone or in combination with another study medicine called sasanlimab at the study clinic.

PF-07921585 will be given as an infusion into a vein or as shots under the skin, once every 3 weeks. Sasanlimab will be given as shots under the skin, also once every 3 weeks.

The experiences of participants receiving the study medicine will be studied to help see if the study medicine is safe and effective. Participants may receive study medicine for up to 2 years, depending on how the cancer responds to the study treatment. Participants may continue receiving study medicine after 2 years if there are any benefits from the study treatment. Participants will attend visits once every 3 weeks with the first 9 weeks having more frequent visits, to check the safety of the study treatment.

DETAILED DESCRIPTION:
The study contains 3 parts:

Part 1: dose escalation of PF-07921585 as single agent to determine the monotherapy recommended dose for further study.

Part 2: dose escalation of PF-07921585 in combination with the anti-PD 1 inhibitor sasanlimab and potentially other anti-cancer agents, in order to determine the recommended dose for expansion of the combination.

Part 3: dose optimization/ expansion will evaluate PF-07921585 in combination with sasanlimab, and potentially other anti-cancer agents. After identification of the recommended dose for expansion in Part 2, participants with select solid tumors will be enrolled into 3-4 cohorts as follows:

* Cohort 1: Melanoma
* Cohort 2: Microsatellite stable (MSS) metastatic colorectal cancer
* Cohort 3: Non-small cell lung cancer (NSCLC)
* Cohort 4: Solid tumor, tumor types and clinical setting to be determined based on emerging data.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants aged ≥18 years or older at the time of informed consent.
2. Tumor types and prior treatment requirements: Participants entering Parts 2 and 3 must have at least 1 measurable lesion.

   Part 1 and Part 2:

   Eligible advanced/metastatic tumor types include NSCLC, urothelial carcinoma (UC), renal cell carcinoma (RCC), melanoma, head and neck squamous cell carcinoma (HNSCC), and microsatellite stable colorectal cancer (MSS-CRC). Participants must have demonstrated radiographic progression on standard treatment(s) for their cancer

   Part 3:
   * Cohort 1: Participants with metastatic melanoma with resistance to checkpoint inhibitor therapy and BRAF/MEKi.
   * Cohort 2: Participants with metastatic MSS-CRC.
   * Cohort 3: Participants with previously untreated metastatic NSCLC.
3. ECOG PS 0 or 1.

Key Exclusion Criteria:

1. Participants with any other active malignancy within 3 years prior to enrollment.
2. Known or suspected hypersensitivity to, or severe allergic history of, human albumin or anti-PD-(L)1 therapy.
3. History of Grade ≥3 immune-related AE (irAE) or unresolved irAEs prior to first dose of study intervention. Exception: vitiligo and endocrinopathy that is controlled with hormonal therapy.
4. History of venous thromboembolic event <12 weeks prior to starting study treatment.
5. Active or history of clinically significant gastrointestinal (GI) disease.
6. Active or history of interstitial lung disease or Grade ≥2 pneumonitis.
7. Active or history of clinically significant autoimmune disease.
8. Active bleeding disorder.
9. Participants who have undergone treatment with any investigational IL-12 agent.
10. Active, uncontrolled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-Limiting Toxicity (DLT) (Parts 1 and 2) | Baseline up to Cycle 2 (each cycle is 21 days)
  Specific adverse events occurring during the first 21 days of study medication and considered at least possibly-related to study medication
Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious AEs (Parts 1 and 2) | Baseline up to 28 days after the last dose of PF-07921585 or after 90 days after the last dose of sasanlimab
  AEs are any untoward medical occurrence in a participant who received study drug. Serious adverse event (SAE) are AEs resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 or 90 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities (Parts 1 and 2) | Baseline up to 28 days after the last dose of PF-07921585 or after 90 days after the last dose of sasanlimab
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Objective Response Rate - Percentage of Participants With Objective Response (Part 3) | Date of first dose up to 2 years
  Percentage of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors 1. 1 (RECIST 1.1).
  CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short aixs was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.

SECONDARY OUTCOMES:
Number of Participants with Treatment emergent Adverse Events (AEs) and Serious AEs (Part 3) | Baseline up to 28 days after the last dose of PF-07921585 and 90 days after the last dose of sasanlimab
  AEs are any untoward medical occurrence in a participant who received study drug. Serious adverse event (SAE) are AEs resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 or 90 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Objective Response Rate-Percentage of Participants with objective response (Parts 1 and 2) | Date of first dose up to 2 years
  Percentage of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors 1. 1 (RECIST 1.1).
  CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short aixs was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Duration of response (DOR)-Parts 1-3 | Date of first dose up to 2 years
  Time in weeks or months from the first documentation of objective tumor response that is subsequently confirmed to objective tumor progression or death due to any cause.
Disease control rate (DCR)-Parts 1-3 | Date of first dose up to 2 years
  DCR is defined as the percent of participants with a confirmed complete response (CR), partial response (PR) or stable disease (SD) according to RECIST 1.1, at 6 weeks.
Progression Free survival (PFS)-Parts 1-3 | Date of first dose until disease progression or death, up to a maximum of 4 years
  Time in weeks or months from first dose to first documentation of objective tumor progression per RECIST 1.1 or death due to any cause.
Overall Survival (OS)-Part 3 | Date of first dose until death, up to a maximum of 4 years
  Time in weeks or months from the start of study treatment to date of death due to any cause.
Pharmacokinetic Parameters: Time to Reach Maximum Observed Plasma Concentration (Tmax)-PF-07921585 | At specific timepoints from Cycle 1 day 1 up to 2 years
  Single dose PK of PF-07921585 as monotherapy (Part 1) and in combination with sansalimab (Parts 2-3) will be calculated. Additional parameters may be calculated if data permits
Pharmacokinetic Parameters: Time to Reach Maximum Observed Plasma Concentration (Tmax ss)-PF-07921585 | At specific timepoints from Cycle 1 day 1 up to 2 years
  Multiple dose PK of PF-07921585 as monotherapy (Part 1) and in combination with sasanlimab (Parts 2-3) will be calculated. Additional parameters may be calculated if data permits
Pharmacokinetic Parameters: Area under the curve (AUCt)-PF-07921585 | At specific timepoints from Cycle 1 day 1 up to 2 years
  Single dose PK of PF-07921585 as monotherapy (Part 1) and in combination with sasanlimab (Parts 2-3) will be calculated. Additional parameters may be calculated if data permits
Pharmacokinetic Parameters: Area under the curve (AUCt ss)-PF-07921585 | At specific timepoints from Cycle 1 day 1 up to 2 years
  Multiple dose PK of PF-07921585 as monotherapy (Part 1) and in combination with sasanlimab (Parts 2-3) will be calculated. Additional parameters may be calculated if data permits
Pharmacokinetic Parameters: Cmax (maximum drug concentration in the body)-PF-07921585 | At specific timepoints from Cycle 1 day 1 up to 2 years
  Single dose PK of PF-07921585 as monotherapy will be calculated. Additional parameters may be calculated if data permits
Pharmacokinetic Parameters: Cmax ss (maximum drug concentration in the body)-PF-07921585 | At specific timepoints from Cycle 1 day 1 up to 2 years
  Multiple dose PK of PF-07921585 as monotherapy (Part 1) and in combination with sasanlimab (Parts 2-3) will be calculated. Additional parameters may be calculated if data permits
Percentage of Participants With Positive PF-07921585 Anti-Drug Antibody (ADA) | At specific timepoints from Cycle 1 day 1 up to 2 years
  Percentage of ADA positive participants by dose level (Parts 1-3)
Percentage of Participants With Positive PF-07921585 neutralizing antibodies (Nab) | At specific timepoints from Cycle 1 Day 1 up to 2 years
  Percentage of Nab positive participants by dose level (Parts 1-3)
Incidence and titer of PF-07921585 ADA and Nab | At specific timepoints from Cycle 1 Day 1 up to 2 years
  Parts 1-3
Pharmacokinetic Parameters: C through-Sasanlimab | At specific timepoints, predose, from Cycle 1 day 1 up to 2 years
  PK of sasanlimab (Parts 2 and 3)
Percentage of Participants With Positive sasanlimab Anti-Drug Antibody (ADA) | At specific timepoints from Cycle 1 day 1 up to 2 years
  Percentage of ADA positive participants by dose level (Parts 2-3)
Percentage of Participants With Positive sasanlimab neutralizing antibodies (Nab) | At specific timepoints from Cycle 1 Day 1 up to 2 years
  Percentage of Nab positive participants by dose level (Parts 2-3)
Incidence and titer of sasanlimab ADA and Nab | At specific timepoints from Cycle 1 Day 1 up to 2 years
  Parts 2-3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Presbyterian/St. Lukes Medical Center, Denver, Colorado
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists Sarasota Drug Development Unit, Sarasota, Florida
  - START Midwest, Grand Rapids, Michigan
  - SCRI Oncology Partners, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5461001